CLINICAL TRIAL: NCT03480802
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Active Comparator-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 Followed by Administration of PNEUMOVAX™23 Eight Weeks Later in Adults Infected With HIV (PNEU-WAY)
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of V114 Followed by PNEUMOVAX™23 in Adults Infected With Human Immunodeficiency Virus (HIV) (V114-018)
Acronym: PNEU-WAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V114-018; V114-018 (Other: Merck Protocol Number); 2017-001909-32 (EudraCT Number)
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Results first posted 2020-11-25 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Pneumococcal Infections
Keywords: Conjugate pneumococcal vaccine, 15-valent, 22F, 33F
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V114 (Experimental): Participants will receive a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2)
  Interventions: Biological: V114; Biological: PNEUMOVAX™23
- Prevnar 13™ (Active Comparator): Participants will receive a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2)
  Interventions: Biological: Prevnar 13™; Biological: PNEUMOVAX™23

INTERVENTIONS:
Biological: V114 — 15-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (2 mcg each), serotype 6B (4 mcg) and Merck Aluminum Phosphate Adjuvant (125 mcg) in each 0.5 mL dose
  Arms: V114
Biological: Prevnar 13™ — 13-valent pneumococcal conjugate vaccine with serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg) and 6B (4.4 mcg) in each 0.5 ml dose
  Arms: Prevnar 13™
Biological: PNEUMOVAX™23 — 23-valent pneumococcal polysaccharide vaccine with serotypes 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19F, 19A, 20, 22F, 23F, 33F (25 mcg each) in each 0.5 mL dose

SUMMARY:
This study is designed to 1) describe the safety, tolerability, and immunogenicity of V114 and Prevnar 13™ in pneumococcal vaccine-naïve adults infected with HIV and to 2) describe the safety, tolerability, and immunogenicity of PNEUMOVAX™23 when administered 8 weeks after receipt of either V114 or Prevnar 13™.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infected with human immunodeficiency virus (HIV) and Cluster of Differentiation 4+ (CD4+) cell count ≥50 cells/µL and plasma HIV ribonucleic acid (RNA) <50,000 copies/mL
* Receiving combination anti-retroviral therapy (ART) for at least 6 weeks before enrollment with no intention of changing therapy for 3 months after randomization
* Female participant: not pregnant, not breastfeeding and 1) not of childbearing potential, or 2) of childbearing potential and agrees to practice contraception through 6 weeks after administration of study vaccine.

Exclusion Criteria:

* History of opportunistic infections within 12 months before the first study vaccination
* History of non-infectious acquired immune deficiency syndrome-related illness such as Kaposi's sarcoma, wasting syndrome, or HIV-associated nephropathy
* History of invasive pneumococcal disease
* Known hypersensitivity to any vaccine component
* Known or suspected congenital immunodeficiency, functional or anatomic asplenia, or history of autoimmune disease
* Coagulation disorder contraindicating intramuscular vaccination
* History of malignancy ≤5 years before enrollment, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Female participant: positive urine or serum pregnancy test
* Prior administration of any pneumococcal vaccine
* Received systemic corticosteroids for ≥14 consecutive days and have not completed within 30 days of enrollment
* Received immunosuppressive therapy
* Received a blood transfusion or blood products within 6 months of enrollment
* Participated in another clinical study of an investigational product within 2 months of enrollment
* Current user of recreational or illicit drugs or recent history of drug or alcohol abuse or dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2018-07-06 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (13):
- United States (4):
  - Bliss Healthcare Services ( Site 0010), Orlando, Florida
  - Triple O Research Institute, P.A. ( Site 0011), West Palm Beach, Florida
  - Saint Hope Foundation, Inc. ( Site 0009), Houston, Texas
  - The Crofoot Research Center, Inc. ( Site 0002), Houston, Texas
- France (3):
  - Hopital Gabriel Montpied ( Site 0084), Clemont Ferrand
  - Hopital Saint Louis ( Site 0094), Paris
  - Hopital Cochin du Paris ( Site 0089), Paris
- Peru (2):
  - Via Libre ( Site 0043), Lima
  - Investigaciones Medicas en Salud - INMENSA ( Site 0041), Lima
- South Africa (2):
  - Chris Hani Baragwanath Hospital ( Site 0122), Johannesburg, Soweto
  - Be Part Yoluntu Centre ( Site 0123), Paarl, Western Cape
- Thailand (2):
  - Siriraj Hosp (Prev&Social Med). ( Site 0183), Bangkok
  - Research Institute for Health. ( Site 0182), Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Mohapi L, Pinedo Y, Osiyemi O, Supparatpinyo K, Ratanasuwan W, Molina JM, Dagan R, Tamms G, Sterling T, Zhang Y, Pedley A, Hartzel J, Kan Y, Hurtado K, Musey L, Simon JK, Buchwald UK; V114-018 (PNEU-WAY) study group. Safety and immunogenicity of V114, a 15-valent pneumococcal conjugate vaccine, in adults living with HIV. AIDS. 2022 Mar 1;36(3):373-382. doi: 10.1097/QAD.0000000000003126. PMID 34750291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults 18 years of age or older infected with human immunodeficiency virus (HIV) who did not receive a pneumococcal vaccine prior to study entry were enrolled in this study.
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2)
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 at Week 8 (Vaccination 2)
Period: Overall Study
Arm/Group | V114 | Prevnar 13™
Started (Vaccinated on Day 1) | 152 | 150
Week 8 (Vaccinated with PNEUMOVAX™23) | 150 | 148
Completed | 145 | 147
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Relocated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 | Prevnar 13™ | Total
Number analyzed (Participants) | 152 | 150 | 302
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.4 (12.5) | 41.3 (12.3) | 41.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 120 | 118 | 238
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 49 | 45 | 94
  Not Hispanic or Latino | 102 | 104 | 206
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 24 | 30 | 54
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 51 | 43 | 94
  White | 41 | 48 | 89
  More than one race | 36 | 26 | 62
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event After Vaccination 1
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs consist of redness/erythema, swelling, and tenderness/pain. The 95% confidence interval (CI) were based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 5 days after Vaccination 1 (Up to Day 5)
Population: All randomized participants who received at least 1 dose of the study vaccination they actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 152 | 150
Percentage of Participants
  Injection site erythema | 4.6 [1.9 to 9.3] | 3.3 [1.1 to 7.6]
  Injection site pain | 57.2 [49.0 to 65.2] | 51.3 [43.0 to 59.6]
  Injection site swelling | 11.8 [7.2 to 18.1] | 4.0 [1.5 to 8.5]

2. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event After Vaccination 1
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited systemic AEs consist of muscle pain (myalgia), joint pain (arthralgia), headache, and tiredness (fatigue). The 95% CI were based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 14 days after Vaccination 1 (Up to Day 14)
Population: All randomized participants who received at least 1 dose of the study vaccination they actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 152 | 150
Percentage of Participants
  Arthralgia | 3.3 [1.1 to 7.5] | 4.0 [1.5 to 8.5]
  Fatigue | 20.4 [14.3 to 27.7] | 13.3 [8.3 to 19.8]
  Headache | 13.2 [8.2 to 19.6] | 9.3 [5.2 to 15.2]
  Myalgia | 12.5 [7.7 to 18.8] | 9.3 [5.2 to 15.2]

3. Primary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event After Vaccination 1
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine is determined by the investigator. The 95% CI were based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Day 1 up to 8 weeks after Vaccination 1 (Up to Week 8)
Population: All randomized participants who received at least 1 dose of the study vaccination they actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 152 | 150
Percentage of Participants | 0 [0.0 to 2.4] | 0 [0.0 to 2.4]

4. Primary Outcome: Geometric Mean Titer (GMT) of Serotype-specific Opsonophagocytic Activity (OPA) After Vaccination 1
Description: Opsonization of pneumococci for phagocytosis is an important mechanism by which antibodies to polysaccharides protect against disease in vivo. Sera from participants was used to measure geometric mean titer (GMT) of 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, using the Multiplexed Opsonophagocytic Assay (MOPA). This assay reads the reciprocal of the highest dilution (1/dil) that gives ≥50% bacterial killing, as determined by comparison to assay background controls. The 95% CIs were derived by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Day 30
Population: All randomized participants without deviations from the protocol that may substantially affect the results of the outcome measure. Deviations include blood draw out of window, prohibited concomitant medication or vaccine, violations of key inclusion/exclusion criteria, or missing serology results.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dil
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 152 | 150
1/dil
  Serotype 1: number analyzed (Participants) | 131 | 131
  Serotype 1 | 238.8 [173.1 to 329.3] | 200.9 [142.7 to 282.7]
  Serotype 3: number analyzed (Participants) | 131 | 130
  Serotype 3 | 116.8 [94.9 to 143.7] | 72.3 [58.6 to 89.2]
  Serotype 4: number analyzed (Participants) | 130 | 131
  Serotype 4 | 824.0 [618.8 to 1097.2] | 1465.5 [1154.5 to 1860.3]
  Serotype 5: number analyzed (Participants) | 131 | 130
  Serotype 5 | 336.7 [242.4 to 467.7] | 276.7 [197.9 to 386.7]
  Serotype 6A: number analyzed (Participants) | 126 | 128
  Serotype 6A | 6421.0 [4890.4 to 8430.7] | 5645.1 [4278.9 to 7447.4]
  Serotype 6B: number analyzed (Participants) | 129 | 130
  Serotype 6B | 4772.9 [3628.3 to 6278.7] | 3554.0 [2751.0 to 4591.4]
  Serotype 7F: number analyzed (Participants) | 131 | 131
  Serotype 7F | 6085.8 [4871.6 to 7602.8] | 6144.3 [4982.8 to 7576.6]
  Serotype 9V: number analyzed (Participants) | 129 | 128
  Serotype 9V | 2836.3 [2311.5 to 3480.4] | 2133.9 [1721.8 to 2644.5]
  Serotype 14: number analyzed (Participants) | 131 | 130
  Serotype 14 | 3508.7 [2730.6 to 4508.5] | 3000.3 [2350.0 to 3830.5]
  Serotype 18C: number analyzed (Participants) | 129 | 129
  Serotype 18C | 3002.2 [2435.5 to 3700.8] | 1560.3 [1213.8 to 2005.6]
  Serotype 19A: number analyzed (Participants) | 131 | 131
  Serotype 19A | 4240.7 [3415.4 to 5265.3] | 3715.9 [2949.2 to 4681.8]
  Serotype 19F: number analyzed (Participants) | 131 | 131
  Serotype 19F | 2438.6 [1972.7 to 3014.6] | 2042.0 [1618.9 to 2575.5]
  Serotype 23F: number analyzed (Participants) | 129 | 127
  Serotype 23F | 1757.4 [1276.1 to 2420.2] | 1787.0 [1309.0 to 2437.9]
  Serotype 22F: number analyzed (Participants) | 128 | 116
  Serotype 22F | 3943.7 [3049.2 to 5100.5] | 109.3 [66.2 to 180.3]
  Serotype 33F: number analyzed (Participants) | 131 | 129
  Serotype 33F | 11342.4 [9184.3 to 14007.6] | 1807.6 [1357.3 to 2407.3]

5. Primary Outcome: Geometric Mean Concentration of Serotype-specific Immunoglobulin G (IgG) After Vaccination 1
Description: The geometric mean concentration of IgG serotype-specific antibodies to the 13 pneumococcal polysaccharide serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) contained in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, were quantitated from participants' sera by multiplex electrochemiluminescence (ECL) using the pneumococcal electrochemiluminescence (PnECL) v2.0 assay, based on the Meso-Scale Discovery technology, which employs disposable multi-spot microtiter plates. The 95% CIs were derived by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Day 30
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 152 | 150
μg/mL
  Serotype 1: number analyzed (Participants) | 139 | 138
  Serotype 1 | 3.16 [2.48 to 4.01] | 4.27 [3.31 to 5.50]
  Serotype 3: number analyzed (Participants) | 139 | 136
  Serotype 3 | 0.57 [0.48 to 0.68] | 0.50 [0.41 to 0.60]
  Serotype 4: number analyzed (Participants) | 138 | 138
  Serotype 4 | 1.14 [0.90 to 1.44] | 2.00 [1.56 to 2.55]
  Serotype 5: number analyzed (Participants) | 139 | 138
  Serotype 5 | 2.38 [1.89 to 3.01] | 2.03 [1.56 to 2.64]
  Serotype 6A: number analyzed (Participants) | 139 | 138
  Serotype 6A | 5.13 [3.73 to 7.04] | 4.91 [3.49 to 6.91]
  Serotype 6B: number analyzed (Participants) | 139 | 138
  Serotype 6B | 7.17 [5.34 to 9.63] | 5.23 [3.73 to 7.35]
  Serotype 7F: number analyzed (Participants) | 139 | 138
  Serotype 7F | 2.61 [2.00 to 3.41] | 3.74 [2.91 to 4.81]
  Serotype 9V: number analyzed (Participants) | 139 | 137
  Serotype 9V | 3.35 [2.71 to 4.14] | 3.55 [2.77 to 4.56]
  Serotype 14: number analyzed (Participants) | 139 | 138
  Serotype 14 | 15.44 [11.69 to 20.39] | 15.22 [11.56 to 20.03]
  Serotype 18C: number analyzed (Participants) | 139 | 138
  Serotype 18C | 5.58 [4.33 to 7.18] | 5.07 [3.97 to 6.48]
  Serotype 19A: number analyzed (Participants) | 139 | 138
  Serotype 19A | 9.09 [7.08 to 11.67] | 9.61 [7.36 to 12.56]
  Serotype 19F: number analyzed (Participants) | 139 | 138
  Serotype 19F | 6.41 [4.89 to 8.39] | 6.21 [4.73 to 8.15]
  Serotype 23F: number analyzed (Participants) | 139 | 138
  Serotype 23F | 3.92 [2.94 to 5.22] | 4.90 [3.54 to 6.77]
  Serotype 22F: number analyzed (Participants) | 139 | 137
  Serotype 22F | 3.97 [3.06 to 5.15] | 0.20 [0.17 to 0.25]
  Serotype 33F: number analyzed (Participants) | 139 | 138
  Serotype 33F | 6.83 [5.14 to 9.07] | 0.77 [0.62 to 0.95]

6. Secondary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event After Vaccination 2
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. Solicited injection-site AEs consist of redness/erythema, swelling, and tenderness/pain. The 95% CI were based on the exact binomial method proposed by Clopper and Pearson.
Time Frame: Up to 5 days after Vaccination 2 (Up to Day 61)
Population: All randomized participants who received at least 1 dose of the study vaccination they actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 150 | 148
Percentage of Participants
  Injection site erythema | 10.0 [5.7 to 16.0] | 12.2 [7.4 to 18.5]
  Injection site pain | 53.3 [45.0 to 61.5] | 61.5 [53.1 to 69.4]
  Injection site swelling | 20.0 [13.9 to 27.3] | 29.1 [21.9 to 37.1]

7. Secondary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event After Vaccination 2
Description: as for outcome 2
Time Frame: Up to 14 days after Vaccination 2 (Up to Day 70)
Population: All randomized participants who received at least 1 dose of the study vaccination they actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 150 | 148
Percentage of Participants
  Arthralgia | 2.7 [0.7 to 6.7] | 1.4 [0.2 to 4.8]
  Fatigue | 12.7 [7.8 to 19.1] | 10.8 [6.3 to 17.0]
  Headache | 8.7 [4.7 to 14.4] | 8.8 [4.8 to 14.6]
  Myalgia | 11.3 [6.7 to 17.5] | 12.2 [7.4 to 18.5]

8. Secondary Outcome: Percentage of Participants With a Vaccine-related Serious Adverse Event After Vaccination 2
Description: as for outcome 3
Time Frame: From Week 8 up to Month 6
Population: All randomized participants who received at least 1 dose of the study vaccination they actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 150 | 148
Percentage of Participants | 0 [0.0 to 2.4] | 0 [0.0 to 2.5]

9. Secondary Outcome: Geometric Mean Titer of Serotype-specific OPA After Vaccination 2
Description: Opsonization of pneumococci for phagocytosis is an important mechanism by which antibodies to polysaccharides protect against disease in vivo. Sera from participants was used to measure GMT of 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) included in V114 and Prevnar 13™; and two serotypes (22F and 33F) which are unique to V114, using the MOPA. The MOPA reads the reciprocal of the highest dilution (1/dil) that gives ≥50% bacterial killing, as determined by comparison to assay background controls. The 95% CIs were derived by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Week 12
Population: All randomized participants without deviations from the protocol that may substantially affect the results of the outcome measure. Deviations include not vaccinated at week 8, vaccination out of window, blood draw out of window, prohibited concomitant medication or vaccine, violations of key inclusion/exclusion criteria, or missing serology results.
Measure: Geometric Mean (95% Confidence Interval); unit: 1/dil
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 150 | 148
1/dil
  Serotype 1: number analyzed (Participants) | 122 | 117
  Serotype 1 | 212.0 [160.5 to 280.2] | 154.0 [111.6 to 212.4]
  Serotype 3: number analyzed (Participants) | 123 | 117
  Serotype 3 | 102.8 [83.0 to 127.2] | 96.6 [79.5 to 117.4]
  Serotype 4: number analyzed (Participants) | 122 | 117
  Serotype 4 | 915.4 [722.9 to 1159.1] | 984.7 [772.1 to 1255.7]
  Serotype 5: number analyzed (Participants) | 123 | 117
  Serotype 5 | 418.1 [312.1 to 560.3] | 274.5 [199.9 to 376.8]
  Serotype 6A: number analyzed (Participants) | 118 | 113
  Serotype 6A | 4065.4 [3052.1 to 5415.1] | 4593.2 [3543.0 to 5954.7]
  Serotype 6B: number analyzed (Participants) | 122 | 117
  Serotype 6B | 3661.1 [2735.1 to 4900.6] | 2826.4 [2202.7 to 3626.8]
  Serotype 7F: number analyzed (Participants) | 122 | 117
  Serotype 7F | 5983.5 [4788.9 to 7476.1] | 5516.5 [4522.2 to 6729.5]
  Serotype 9V: number analyzed (Participants) | 120 | 117
  Serotype 9V | 2454.8 [2008.7 to 3000.0] | 1929.9 [1567.7 to 2375.7]
  Serotype 14: number analyzed (Participants) | 123 | 117
  Serotype 14 | 3634.0 [2935.6 to 4498.5] | 2539.3 [1960.6 to 3288.9]
  Serotype 18C: number analyzed (Participants) | 122 | 115
  Serotype 18C | 2511.5 [1958.7 to 3220.3] | 1753.8 [1428.6 to 2153.1]
  Serotype 19A: number analyzed (Participants) | 123 | 117
  Serotype 19A | 3358.1 [2679.6 to 4208.4] | 3300.3 [2638.7 to 4127.7]
  Serotype 19F: number analyzed (Participants) | 123 | 116
  Serotype 19F | 2230.7 [1803.6 to 2759.0] | 1994.1 [1630.7 to 2438.4]
  Serotype 23F: number analyzed (Participants) | 120 | 116
  Serotype 23F | 1641.2 [1217.2 to 2212.9] | 1266.5 [944.3 to 1698.5]
  Serotype 22F: number analyzed (Participants) | 121 | 116
  Serotype 22F | 3399.9 [2697.6 to 4285.0] | 2952.7 [2207.7 to 3949.1]
  Serotype 33F: number analyzed (Participants) | 123 | 117
  Serotype 33F | 10576.3 [8383.1 to 13343.4] | 11926.3 [9085.9 to 15654.6]

10. Secondary Outcome: Geometric Mean Concentration of Serotype-specific IgG After Vaccination 2
Description: The geometric mean concentration of IgG serotype-specific antibodies to the 13 pneumococcal polysaccharide serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) contained in V114 and Prevnar 13™ ; and two serotypes (22F and 33F) which are unique to V114, were quantitated from participants' sera by multiplex ECL using the PnECL v2.0 assay, based on the Meso-Scale Discovery technology, which employs disposable multi-spot microtiter plates. The 95% CIs were derived by exponentiating the CIs of the mean of the natural log values based on the t-distribution.
Time Frame: Week 12
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V114 | Prevnar 13™
Number analyzed (Participants) | 150 | 148
μg/mL
  Serotype 1: number analyzed (Participants) | 130 | 129
  Serotype 1 | 2.80 [2.25 to 3.49] | 4.04 [3.27 to 5.00]
  Serotype 3: number analyzed (Participants) | 130 | 128
  Serotype 3 | 0.51 [0.43 to 0.61] | 0.59 [0.50 to 0.70]
  Serotype 4: number analyzed (Participants) | 130 | 129
  Serotype 4 | 1.26 [1.10 to 1.57] | 1.61 [1.31 to 1.98]
  Serotype 5: number analyzed (Participants) | 130 | 129
  Serotype 5 | 2.61 [2.08 to 3.28] | 2.13 [1.69 to 2.68]
  Serotype 6A: number analyzed (Participants) | 130 | 129
  Serotype 6A | 3.12 [2.27 to 4.30] | 3.71 [2.74 to 5.03]
  Serotype 6B: number analyzed (Participants) | 130 | 129
  Serotype 6B | 4.69 [3.52 to 6.25] | 4.35 [3.23 to 5.86]
  Serotype 7F: number analyzed (Participants) | 130 | 129
  Serotype 7F | 2.45 [1.91 to 3.15] | 3.17 [2.60 to 3.87]
  Serotype 9V: number analyzed (Participants) | 130 | 128
  Serotype 9V | 2.92 [2.39 to 3.57] | 3.24 [2.62 to 4.01]
  Serotype 14: number analyzed (Participants) | 130 | 129
  Serotype 14 | 13.68 [10.34 to 18.10] | 14.37 [11.25 to 18.36]
  Serotype 18C: number analyzed (Participants) | 130 | 129
  Serotype 18C | 3.96 [3.08 to 5.09] | 3.96 [3.18 to 4.95]
  Serotype 19A: number analyzed (Participants) | 130 | 129
  Serotype 19A | 7.23 [5.80 to 9.02] | 8.54 [6.80 to 10.72]
  Serotype 19F: number analyzed (Participants) | 130 | 129
  Serotype 19F | 5.19 [4.06 to 6.62] | 5.84 [4.67 to 7.30]
  Serotype 23F: number analyzed (Participants) | 130 | 129
  Serotype 23F | 3.21 [2.42 to 4.25] | 3.74 [2.85 to 4.91]
  Serotype 22F: number analyzed (Participants) | 130 | 129
  Serotype 22F | 3.94 [3.07 to 5.05] | 3.50 [2.75 to 4.45]
  Serotype 33F: number analyzed (Participants) | 130 | 129
  Serotype 33F | 6.18 [4.72 to 8.09] | 9.20 [7.19 to 11.77]

ADVERSE EVENTS:
Time Frame: V114 and Prevnar 13™ arms: NSAEs from Day 1 up to 14 days after vaccination 1, and SAEs from Day 1 up to Week 8. V114 (Post-PPV23) and Prevnar 13™ (Post-PPV23) arms: NSAEs from week 8 up to 14 days after vaccination 2, and SAEs after Week 8 vaccination up to Month 6. All-Cause Mortality: From screening up to Month 6.
Description: The population reported was all randomized participants who received study intervention at the specified timepoint. Adverse events were reported (1) following administration of either V114 or Prevnar 13™ and (2) following administration of PNEUMOVAX™23 (PPV23).
Groups:
- V114: Participants received a single 0.5 mL intramuscular (IM) injection of V114 on Day 1 (Vaccination 1).
- Prevnar 13™: Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1).
- V114 (Post-PPV23): Participants received a single 0.5 mL IM injection of V114 on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PNEUMOVAX™23 (PPV23) at Week 8 (Vaccination 2).
- Prevnar 13™ (Post-PPV23): Participants received a single 0.5 mL IM injection of Prevnar 13™ on Day 1 (Vaccination 1) and a single 0.5 mL IM injection of PPV23 at Week 8 (Vaccination 2).
Arm/Group | V114 | Prevnar 13™ | V114 (Post-PPV23) | Prevnar 13™ (Post-PPV23)
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/150 | 0/150 | 0/148
Serious Adverse Events (participants affected / at risk) | 3/152 | 0/150 | 2/150 | 6/148
Other Adverse Events (participants affected / at risk) | 103/152 | 88/150 | 88/150 | 99/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=152) | Prevnar 13™ (N=150) | V114 (Post-PPV23) (N=150) | Prevnar 13™ (Post-PPV23) (N=148)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 (N=152) | Prevnar 13™ (N=150) | V114 (Post-PPV23) (N=150) | Prevnar 13™ (Post-PPV23) (N=148)
Fatigue (General disorders) | 31 (34) | 20 (23) | 19 (20) | 16 (16)
Injection site erythema (General disorders) | 8 (8) | 5 (5) | 15 (15) | 18 (18)
Injection site pain (General disorders) | 88 (100) | 78 (86) | 80 (97) | 92 (101)
Injection site swelling (General disorders) | 18 (18) | 6 (6) | 30 (30) | 43 (43)
Myalgia (Musculoskeletal and connective tissue disorders) | 19 (21) | 14 (15) | 17 (18) | 18 (18)
Headache (Nervous system disorders) | 20 (23) | 14 (15) | 13 (14) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT03480802/Prot_SAP_000.pdf